CLINICAL TRIAL: NCT03886883
Title: Endogenous Modulation of Pain - the Tolerance to Stretch
Brief Title: Endogenous Modulation of Pain and Stretch Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UniversityCND1
Record Dates: First submitted 2019-03-13; First posted 2019-03-22 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Pain Threshold
Keywords: Stretch tolerance; Stretching Exercises; Exercise induced hypoalgesia
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: This was a randomized, repeated-measures cross-over study. Passive knee extension range of motion was measured three consecutive times with five-minute intervals between measurements. Both groups underwent a static stretch protocol consisting of two bouts of thirty-second constant-angle static stretching of the knee flexors with a one-minute rest between bouts. Subjects were instructed to keep the limb relaxed as the lower leg was passively moved towards extension. Following stretching, the post-stretch measurement was performed. Finally, subjects in the pain group were instructed to immerse their non-dominant hand into a container with circulating water at 1˚C to 4˚C and keep it there for 2 minutes. A Biodex system 4 pro dynamometer was used to quantify range of motion and passive resistive torque. Pressure pain thresholds was assessed using a handheld pressure algometer (Somedic AB, Hörby, Sweden).
Who Masked: Participant
Masking Description: Participants were blinded to the results of all measurements and naïve to research hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise-induced hypoalgesia (EIH) (Experimental): Exercise-induced hypoalgesia - isometric muscle contractions of the hand flexors
  Interventions: Other: Exercise induced hypoalgesia (EIH)
- Static stretch (SS) (Active Comparator): A static stretch of the knee flexors
  Interventions: Other: Static stretch (SS)
- Rest (Sham Comparator): No intervention
  Interventions: Other: Rest
- Conditioning painful stimulus (CPM) (Experimental): Conditioned pain modulation - cold pressure test
  Interventions: Other: Conditioned pain modulation (CPM)

INTERVENTIONS:
Other: Exercise induced hypoalgesia (EIH) — An EIH response was induced by a 3-minute isometric contraction of the hand flexor muscles at 25% of maximal voluntary contraction (MVC).
  Arms: Exercise-induced hypoalgesia (EIH)
Other: Static stretch (SS) — Two bouts of 30 seconds of static stretching (SS) of the knee flexors.
  Arms: Static stretch (SS)
Other: Rest — The participants rested in a seated position for 10 minutes
  Arms: Rest
Other: Conditioned pain modulation (CPM) — A CPM response was induced by way of the cold pressor test.
  Arms: Conditioning painful stimulus (CPM)

SUMMARY:
This study investigates the role of two endogenous inhibitory mechanisms; exercise-induced hypoalgesia (EIH) and a conditioning painful stimulus (CPM) on passive joint range of motion, passive resistive torque and pain sensitivity. The study is a randomized, repeated-measures cross-over study.

DETAILED DESCRIPTION:
The increase in range of motion following stretching is related to changes in the tolerance to stretch. The mechanistic relationships behind these changes in subject sensation are however unknown but could be related to endogenous modulation of pain.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for participation included the absence of any pain or other conditions that might affect the somatosensory system.

Exclusion Criteria:

* Substance abuse, History of neurological or mental disabilities, Lack of ability to comply with instructions, Delayed onset of muscle soreness.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only males were included to avoid the potential effect that fluctuations in gonadal hormone values may have on the endogenous pain inhibitory mechanisms.
Enrollment: 19 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Knee extension range of motion | Passive knee extension range of motion was measured as a baseline just prior to the induction of exercise-induced hypoalgesia (EIH), Static stretch (SS), Rest and a conditioning painful stimulus (CPM)
  Passively induced knee extension range of motion was measured using the Biodex system 4 pro isokinetic dynamometer
Knee extension range of motion | Passive knee extension range of motion was measured 30 seconds after the induction of EIH, SS, Rest and CPM
  Passively induced knee extension range of motion was measured using the Biodex system 4 pro isokinetic dynamometer
Knee extension range of motion | Passive knee extension range of motion was measured 10 minutes after the induction of EIH, SS, Rest and CPM
  Passively induced knee extension range of motion was measured using the Biodex system 4 pro isokinetic dynamometer

SECONDARY OUTCOMES:
Passive resistive torque | Passive resistive torque was measured as a baseline just prior to the induction of EIH, SS, Rest and CPM
  Passive resistive torque during the passive knee extension motion was measured using the Biodex system 4 pro isokinetic dynamometer.
Passive resistive torque | Passive resistive torque was measured 30 seconds after the induction of EIH, SS, Rest and CPM
  Passive resistive torque during the passive knee extension motion was measured using the Biodex system 4 pro isokinetic dynamometer.
Passive resistive torque | Passive resistive torque was measured 10 minutes after the induction of EIH, SS, Rest and CPM
  Passive resistive torque during the passive knee extension motion was measured using the Biodex system 4 pro isokinetic dynamometer.
Pressure pain thresholds | Pressure pain thresholds were measured as a baseline just prior to the induction of EIH, SS, Rest and CPM
  Pressure pain thresholds was measures using a handheld pressure algometer (Somedic AB, Hörby, Sweden.
Pressure pain thresholds | Pressure pain thresholds were measured 30 seconds after the induction of EIH, SS, Rest and CPM
  Pressure pain thresholds was measures using a handheld pressure algometer (Somedic AB, Hörby, Sweden.
Pressure pain thresholds | Pressure pain thresholds were measured 10 minutes after the induction of EIH, SS, Rest and CPM
  PRessure pain thresholds was measures using a handheld pressure algometer (Somedic AB, Hörby, Sweden.

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Drachman, Msc., Study Director — University College of Northern Denmark, Department of Physiotherapy
Locations (1):
- University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stove MP, Hirata RP, Palsson TS. The tolerance to stretch is linked with endogenous modulation of pain. Scand J Pain. 2021 Jan 11;21(2):355-363. doi: 10.1515/sjpain-2020-0010. Print 2021 Apr 27. PMID 34387949